CLINICAL TRIAL: NCT06087952
Title: Leiden Thrombosis Recurrence Risk Prevention: Tailored Treatment After a First Venous Thromboembolism
Brief Title: Leiden Thrombosis Recurrence Risk Prevention
Acronym: L-TRRiP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Suzanne C. Cannegieter, MD PhD, Professor of Clinical Epidemiology, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P20.090; 848017007 (Other Grant/Funding Number: ZonMw the Netherlands); NL74711.058.20 (Other: ToetsingOnline); NL9003 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2023-07-25; First posted 2023-10-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboembolism; Venous Thromboses; Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients with low recurrent VTE risk are advised to stop anticoagulant therapy. Patients with high recurrent VTE risk and low bleeding risk are advised to continue anticoagulant therapy.
  Patients with intermediate recurrent VTE risk, or high recurrent VTE risk and high bleeding risk are randomised to stop or continue anticoagulant therapy.
Masking Description: Blinded endpoint adjudication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Continue anticoagulation (Other): Patients with high recurrent VTE risk and low major bleeding risks are advised to continue anticoagulant therapy.
  Interventions: Diagnostic Test: VTE-BLEED score; Diagnostic Test: L-TRRiP score; Other: Advise to continue anticoagulant treatment after 3 months
- Discontinue anticoagulation (Other): Patients with low recurrent VTE risk are advised to discontinue anticoagulant therapy.
  Interventions: Diagnostic Test: VTE-BLEED score; Diagnostic Test: L-TRRiP score; Other: Advise to discontinue anticoagulant treatment after 3 months
- Randomised to continue anticoagulation (Other): Patients with intermediate recurrent VTE risk or high recurrent VTE risk and high major bleeding risk are randomised to continue or discontinue anticoagulant therapy.
  Interventions: Other: Randomised treatment advice (discontinue vs continue after 3 months); Diagnostic Test: VTE-BLEED score; Diagnostic Test: L-TRRiP score
- Randomised to discontinue anticoagulation (Other): Patients with intermediate recurrent VTE risk or high recurrent VTE risk and high major bleeding risk are randomised to continue or discontinue anticoagulant therapy.
  Interventions: Other: Randomised treatment advice (discontinue vs continue after 3 months); Diagnostic Test: VTE-BLEED score; Diagnostic Test: L-TRRiP score

INTERVENTIONS:
Other: Randomised treatment advice (discontinue vs continue after 3 months) — Randomisation to continue or discontinue anticoagulant therapy in 1:1 ratio stratified on risk category of L-TRRiP and VTE-BLEED score
  Arms: Randomised to continue anticoagulation; Randomised to discontinue anticoagulation
Diagnostic Test: VTE-BLEED score — Predict bleeding risk during extended anticoagulant treatment (high or low) using the VTE-BLEED score
Diagnostic Test: L-TRRiP score — Predict VTE recurrence risk after anticoagulant discontinuation (high, intermediate or low) using the L-TRRiP score
Other: Advise to continue anticoagulant treatment after 3 months — Advise to continue anticoagulant treatment after 3 months for patients with high VTE recurrence and low bleeding risk
  Arms: Continue anticoagulation
Other: Advise to discontinue anticoagulant treatment after 3 months — Advise to discontinue anticoagulant treatment after 3 months for patients with low VTE recurrence risk
  Arms: Discontinue anticoagulation

SUMMARY:
The goal of this clinical trial is to evaluate tailored duration of long-term anticoagulant treatment after a first venous thromboembolism based on individualized risk assessments of recurrent VTE and major bleeding risks.

Participants will be asked to fill in a questionnaire and take a buccal swab, which are used for an individual estimation of the risks of recurrent VTE and bleeding. Based on these risks a treatment advise will be made, or randomised in a subgroup of patients.

DETAILED DESCRIPTION:
Background: Patients with a first venous thromboembolism (VTE) are at risk of recurrence. A recurrent VTE can be prevented by prolonged anticoagulant therapy, but this may come at the cost of major bleeding. The L-TRRiP and VTE-BLEED prediction scores have been developed to classify the risk of recurrent VTE (low, intermediate, high) and major bleeding (low vs high), respectively. However, their combined use in finding the optimal balance to minimize both long-term risks is unclear.

Aims: To evaluate tailored duration of long-term anticoagulant treatment based on individualized risk assessments of recurrent VTE and major bleeding risks.

Methods:

The L-TRRiP study is a multicenter, open-label, cohort based randomized controlled trial in which patients with a first VTE will be included. For each patient the risk of recurrent VTE (low, medium, high) and major bleeding (low, high) will be determined using the L-TRRiP and VTE-BLEED prediction scores, respectively. After three months of initial anticoagulant therapy, patients with a low recurrent VTE risk (<6% in 2 years) will discontinue anticoagulants, whereas patients with a high recurrent VTE risk(>14% in 2 years) and low major bleeding risk will continue. The other groups, with unclear benefit of prolonged treatment, will be randomized to continue or discontinue anticoagulants. Patients will be followed for at least two years, during which they will be asked to fill in a questionnaire every 3 months during the first two years, followed by a questionnaire once a year for the remaining duration of the study (i.e., 2 years after inclusion of the last participant; which is expected to be in 2027). The total follow-up duration is therefore expected to vary between 2 to 6 years. The follow-up questionnaires are used to screen for potential outcomes (including recurrent VTE and bleeding), and includes the EQ-5D-5L to assess quality of life, the Post VTE functional status scale to assess functional outcomes and the Medical Consumption and Productivity Costs Questionnaire to asses cost-effectiveness. In case of a potential outcome additional information is retrieved from the medical record for adjudication. The clinical outcomes will be evaluated and classified by an independent committee blinded for treatment allocation.

Sample size: The sample size of this study is based on the randomized part of the study. To demonstrate a 7% difference in the combined endpoint (i.e., 10.6% vs 3.6%) with an alpha of 0.05 and a power of 90%, a sample size of 552 subjects for the randomized part of the study is required. Taking into account a drop-out rate of 10%, the aim is to include 608 patients in the randomized part of the study. After inclusion of 608 randomized patients, inclusion will stop. Based on the derivation studies it is expected the randomized group will form about 40% of the total included population, in which case the estimated total number of included patients will be 1600. Of note, this total number may change depending on the final proportion of the randomized group.

Ethics: The study has been approved by the Medical Ethics Committee Leiden Den Haag Delft. All participants will provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Be diagnosed with a first confirmed symptomatic deep vein thrombosis (including distal vein thrombosis, in Dutch: 'kuitvenetrombose') or pulmonary embolism with an indication for treatment with anticoagulant therapy for at least 3 months as prescribed by their treating physician.
3. Be aged 18 years or above.

Exclusion Criteria:

1. Patients with active cancer (i.e. cancer diagnosis within six months before VTE (excluding basal-cell or squamous-cell carcinoma of the skin), recently recurrent or progressive cancer or any cancer that required anti-cancer treatment within six months before the venous thromboembolism was diagnosed) or antiphospholipid syndrome
2. Patients who need to continue anticoagulant treatment for another indication (e.g. atrial fibrillation).
3. Patients with a strong indication for long-term antiplatelet therapy despite oral anticoagulation (e.g. those with recent STEMI)
4. Patients with COVID-19 associated VTE (hospital admission because of COVID-19 <3 months before the VTE) or vaccine-induced immune thrombotic thrombocytopenia (VITT)
5. Patients in whom the risk of bleeding is deemed extremely high by the treating physician, necessitating discontinuation of anticoagulant treatment for the first VTE after the initial 3 months or even during the initial 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent VTE and major bleeding | 2 years
  Incidence of the combined endpoint recurrent VTE and major bleeding in the randomised arms

SECONDARY OUTCOMES:
Primary outcome weighted for quality of life (EQ-5D-5L) | 2 years
  Recurrent VTE and major bleeding weighted for the impact on quality of life as measured by the EQ-5D-5L
Primary outcome weighted for functional status (PFVS) | 2 years
  Recurrent VTE and major bleeding weighted for the impact on functional limitations as measured by the Post-VTE functional status scale (PFVS) a grade for functional outcomes after a VTE, ranging from grade 0 (no functional limitations, symptoms, pain or anxiety) to grade 4 (severe functional limitations, requiring assistance in activities of daily living) or death..
Cost-effectiveness | Up to 2 years
  For the analysis of cost-effectiveness health care costs and productivity losses will be measured every 3 months during follow-up by the Medical Consumption Questionnaire and Productivity Costs Questionnaire from the institute for Medical Technology Assessment. Health care costs will be calculated using Dutch standard prices for economic evaluations. Absence from work will be valued with friction cost method. Quality Adjusted Life Years (QALYs) will be assessed using the EQ-5D-5L score, which is taken every 3 months during follow-up, using the area-under-the-curve approach. Economic evaluation will consists of both a study-based cost-effectiveness analysis (cost per event) as well as cost-utility analysis with a lifetime horizon (costs per QALY).
Recurrent VTE and major bleeding in non-randomised arms | 2 years
  Incidence of the combined endpoint in the non-randomised arms
Clinically relevant non-major bleeding | 2 years
  Incidence of clinically relevant non-major bleeding in different study arms
Reccurent VTE, major bleeding and clinically relevant - non Major bleeding during entire follow-up | Up to 6 years
  Incidence of recurrent VTE, major bleeding and clinically relevant bleeding in different study arms for the entire duration of follow-up (expected to vary between 2 to 6 years)
Predictive performance of the L-TRRiP model | Up to 6 years
  Discrimination and calibration of L-TRRiP model in the arms that discontinue anticoagulant treatment
Predictive performance of the VTE-BLEED model | Up to 6 years
  Discrimination and calibration of the L-TRRiP model in the arms that continue anticoagulant treatment
Natural course of recovery | Up to 6 years
  Natural course of recovery with regard to long-term functional limitations, measured by post VTE functional status scale every 3 months through the follow-up period of 2 years. Using the post VTE functional status scale (PFVS) a grade for functional outcomes after a VTE, ranging from grade 0 (no functional limitations, symptoms, pain or anxiety) to grade 4 (severe functional limitations, requiring assistance in activities of daily living) or death.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Cannegieter, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (19):
- Netherlands (19):
  - Leiden University Medical Center, Leiden, South Holland
  - Amsterdam Medical Center, location AMC, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Nij Smellinghe Ziekenhuis, Drachten
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - HagaZiekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
After data collection and data cleaning are finished deidentified data will be registered in a repository and be made available for further research upon reasonable request to the corresponding author.

REFERENCES:
- [Derived] Burggraaf-van Delft JLI, van Rein N, Bemelmans RHH, van den Berg JK, Bruggeman CY, Cloos-van Balen M, Coppens M, Eefting M, Ende-Verhaar Y, van Es N, van Guldener C, de Jong WK, Kleijwegt F, Koster T, Kroon C, Kuipers S, Leentjens J, Luijten D, Mairuhu ATA, Meijer K, van de Ree MA, Roos R, Schrover I, Swart-Heikens J, van der Velden AWG, van den Akker-van Marle EM, le Cessie S, Geersing GJ, Middeldorp S, Huisman MV, Klok FA, Cannegieter SC; L-TRRiP investigators. Tailored anticoagulant treatment after a first venous thromboembolism: protocol of the Leiden Thrombosis Recurrence Risk Prevention (L-TRRiP) study - cohort-based randomised controlled trial. BMJ Open. 2024 Mar 23;14(3):e078676. doi: 10.1136/bmjopen-2023-078676. PMID 38521524